CLINICAL TRIAL: NCT01068600
Title: A 12-week Treatment, Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Assess the Efficacy and Safety of Once Daily Indacaterol in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Comparison of Efficacy of Indacaterol Versus Placebo Over 12 Weeks
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQAB149B2355
Record Dates: First submitted 2010-02-12; First posted 2010-02-15 (Estimated); Results first posted 2011-08-19 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Indacaterol
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Indacaterol 75 µg (Experimental): Indacaterol 75 µg inhaled once daily in the morning via Concept1, a single dose dry powder inhaler (SDDPI), for 12 weeks.
  Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol
- Placebo (Placebo Comparator): Placebo to indacaterol inhaled once daily in the morning via Concept1, a SDDPI, for 12 weeks.
  Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) albuterol was available for rescue use throughout the study.
  Interventions: Drug: Placebo to indacaterol

INTERVENTIONS:
Drug: Indacaterol — Once daily via single-dose dry powder inhaler (SDDPI)
  Arms: Indacaterol 75 µg
Drug: Placebo to indacaterol — Once daily via SDDPI
  Arms: Placebo

SUMMARY:
This 12-week study evaluated the efficacy and safety of indacaterol versus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD (moderate-to-severe as classified by the Global Initiative for Chronic Obstructive Lung Disease (GOLD) Guidelines, 2008) and:

  1. Smoking history of at least 10 pack-years
  2. Post-bronchodilator FEV1 <80% and ≥30% of the predicted normal value
  3. Post-bronchodilator FEV1/FVC (forced vital capacity) <70%

Exclusion Criteria:

* Patients who have had a COPD exacerbation requiring systemic corticosteroids and/or antibiotics and/or hospitalization for in the 6 weeks prior to screening
* Patients who have had a respiratory tract infection within 6 weeks prior to screening
* Patients with concomitant pulmonary disease
* Patients with a history of asthma
* Patients with diabetes Type I or uncontrolled diabetes Type II
* Any patient with lung cancer or a history of lung cancer
* Patients with a history of certain cardiovascular comorbid conditions

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (49):
- United States (49):
  - Novartis Investigative Site, Anniston, Alabama
  - Novartis Investigative Site, Jasper, Alabama
  - Novartis Investigator Site, Glendale, Arizona
  - Novartis Investigator Site, Phoenix, Arizona
  - Novartis Investigator Site, Fullerton, California
  - Novartis Investigator Site, Los Angeles, California
  - Novartis Investigator Site, Riverside, California
  - Novartis Investigative Site, Clearwater, Florida
  - Novartis Investigative Site, Hollywood, Florida
  - Novartis Investigative site, Miami, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Winter Park, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigator Site, Normal, Illinois
  - Novartis Investigator Site, Iowa City, Iowa
  - Novartis Investigative Site, Madisonville, Kentucky
  - Novartis Investigator Site, Baton Rouge, Louisiana
  - Novartis Investigator Site, Opelousas, Louisiana
  - Novartis Investigator Site, Saint Charles, Missouri
  - Novartis Investigator Site, St Louis, Missouri
  - Novartis Investigator Site, Lincoln, Nebraska
  - Novartis Investigator Site, Omaha, Nebraska
  - Novartis Investigator Site, Henderson, Nevada
  - Novartis Investigator Site, Las Vegas, Nevada
  - Novartis Investigative Site, Cherry Hill, New Jersey
  - Novartis Investigator Site, Albuquerque, New Mexico
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigative Site, Shelby, North Carolina
  - Novartis Investigative Site, Canton, Ohio
  - Novartis Investigator Site, Cincinnati, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigator Site, Marion, Ohio
  - Novartis Investigator Site, Eugene, Oregon
  - Novartis Investigator Site, Medford, Oregon
  - Novartis Investigative Site, Cumberland, Rhode Island
  - Novartis Investigative Site, Pawtucket, Rhode Island
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Easley, South Carolina
  - Novartis Investigative site, Greenville, South Carolina
  - Novartis Investigative Site, North Charleston, South Carolina
  - Novartis Investigative Site, Spartanburg, South Carolina
  - Novartis Investigative Site, Union, South Carolina
  - Novartis Investigator Site, Arlington, Texas
  - Novartis Investigator Site, Dickinson, Texas
  - Novartis Investigator Site, El Paso, Texas
  - Novartis Investigator Site, McKinney, Texas
  - Novartis Investigative Site, South Burlington, Vermont
  - Novartis Investigative Site, Richmond, Virginia

REFERENCES:
- [Derived] Gotfried MH, Kerwin EM, Lawrence D, Lassen C, Kramer B. Efficacy of indacaterol 75 mug once-daily on dyspnea and health status: results of two double-blind, placebo-controlled 12-week studies. COPD. 2012 Dec;9(6):629-36. doi: 10.3109/15412555.2012.729623. Epub 2012 Sep 28. PMID 23020650
- [Derived] Kerwin EM, Gotfried MH, Lawrence D, Lassen C, Kramer B. Efficacy and tolerability of indacaterol 75 mug once daily in patients aged >/=40 years with chronic obstructive pulmonary disease: results from 2 double-blind, placebo-controlled 12-week studies. Clin Ther. 2011 Dec;33(12):1974-84. doi: 10.1016/j.clinthera.2011.11.009. PMID 22177371

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Indacaterol 75 µg | Placebo
Started | 159 | 159
Completed | 148 | 142
Not Completed | 11 | 17
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Adverse Event | 3 | 3
Not completed — Abnormal laboratory value(s) | 1 | 0
Not completed — Lost to Follow-up | 1 | 2
Not completed — Protocol deviation | 1 | 1
Not completed — Unsatisfactory therapeutic effect | 0 | 4
Not completed — Administrative problems | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indacaterol 75 µg | Placebo | Total
Number analyzed (Participants) | 159 | 159 | 318
Age Continuous [Mean (Standard Deviation); unit: years] | 61.3 (9.83) | 61.5 (9.85) | 61.4 (9.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 70 | 146
  Male | 83 | 89 | 172

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) After 12 Weeks of Treatment
Description: Spirometry was conducted according to internationally accepted standards. Trough FEV1 was defined as the average of the 23 hour 10 minute and 23 hour 45 minute post-dose FEV1 readings. Mixed model used baseline FEV1, FEV1 prior to and 10-15 minutes post inhalation of albuterol, and FEV1 prior to and 50-70 minutes post inhalation of ipratropium as covariates.
Time Frame: after 12 weeks
Population: Full Analysis Set included all randomized participants who received at least one dose of study drug. The endpoint was analyzed only for those participants who had data for this outcome measure. Missing data was imputed using last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 75 µg | Placebo
Number analyzed (Participants) | 145 | 150
Liters | 1.49 (0.016) | 1.35 (0.015)

2. Secondary Outcome: Transition Dyspnoea Index (TDI) Focal Score After 12 Weeks of Treatment
Description: TDI focal score is based on three domains: functional impairment, magnitude of task and magnitude of effort. Each domain is scored from -3 (major deterioration) to 3 (major improvement) to give an overall TDI focal score of -9 to 9 with a negative score indicating a deterioration from baseline. A 1 unit difference in the TDI focal score is clinically significant. Mixed model used baseline dyspnoea index, FEV1 prior to and 10-15 minutes post inhalation of albuterol, and FEV1 prior to and 50-70 minutes post inhalation of ipratropium as covariates.
Time Frame: after 12 weeks
Population: Full Analysis Set included all randomized participants who received at least one dose of study medication. If data were missing or insufficient for any one of the domains a focal score was not calculated. Missing focal scores after week 4 were imputed using last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Indacaterol 75 µg | Placebo
Number analyzed (Participants) | 148 | 149
Score on a scale | 1.22 (0.234) | 0.76 (0.235)

ADVERSE EVENTS:
Description: Safety set included all randomized participants who received study drug.
Arm/Group | Indacaterol 75 µg | Placebo
Serious Adverse Events (participants affected / at risk) | 4/159 | 4/159
Other Adverse Events (participants affected / at risk) | 58/159 | 46/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 75 µg (N=159) | Placebo (N=159)
Splenic infarction (Blood and lymphatic system disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 75 µg (N=159) | Placebo (N=159)
Supraventricular extrasystoles (Cardiac disorders) | 2 | 0
Ear pain (Ear and labyrinth disorders) | 2 | 0
Vision blurred (Eye disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 2 | 0
Oedema peripheral (General disorders) | 2 | 1
Seasonal allergy (Immune system disorders) | 2 | 0
Bronchitis (Infections and infestations) | 4 | 2
Lower respiratory tract infection (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 10 | 3
Pneumonia (Infections and infestations) | 2 | 2
Sinusitis (Infections and infestations) | 1 | 6
Upper respiratory tract infection (Infections and infestations) | 5 | 6
Upper respiratory tract infection bacterial (Infections and infestations) | 3 | 2
Urinary tract infection (Infections and infestations) | 1 | 4
Viral upper respiratory tract infection (Infections and infestations) | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 2
Blood creatine phosphokinase increased (Investigations) | 1 | 3
C-reactive protein increased (Investigations) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Headache (Nervous system disorders) | 5 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 13 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Hypertension (Vascular disorders) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.